CLINICAL TRIAL: NCT03234478
Title: Parkinson Disease and DBS: Cognitive Effects in GBA Mutation Carriers
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Gian Dev Pal, MD, MS, Assistant Professor of Neurological Sciences, Rutgers, The State University of New Jersey
Other Study IDs: Pro2020000729; 1K23NS097625-01A1 (NIH)
Record Dates: First submitted 2017-07-25; First posted 2017-07-31 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Parkinson; Parkinson Disease; Genetic Predisposition; GBA Gene Mutation; Cognitive Decline
Keywords: deep brain stimulation; cognition; young onset Parkinson disease
MeSH Terms: conditions — Parkinson Disease; Genetic Predisposition to Disease; Cognitive Dysfunction; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood will be retained for analysis of GBA metabolites.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- GBA mutation carriers without DBS: Parkinson's disease patients who have moderate to advanced disease but have not undergone deep brain stimulation. Subjects will be tested for GBA mutation status as part of this study.
  Interventions: Other: cognitive assessments
- non-mutation carriers without DBS: Parkinson's disease patients who have moderate to advanced disease but have not undergone deep brain stimulation. Subjects will be tested for GBA mutation status as part of this study.
  Interventions: Other: cognitive assessments
- GBA mutation carriers with DBS: Parkinson's disease patients who have moderate to advanced disease and have undergone deep brain stimulation. Subjects will be tested for GBA mutation status as part of this study.
  Interventions: Other: cognitive assessments
- non-mutation carriers with DBS: Parkinson's disease patients who have moderate to advanced disease and have undergone deep brain stimulation. Subjects will be tested for GBA mutation status as part of this study.
  Interventions: Other: cognitive assessments

INTERVENTIONS:
Other: cognitive assessments — Cognitive assessments will be performed at baseline, 1 year, and 2 years, depending on subject cohort placement

SUMMARY:
Every year, approximately 9,000 Parkinson disease (PD) patients undergo deep brain stimulator (DBS) placement into the subthalamic nucleus (STN-DBS). Studies suggest that PD patients with mutations in the glucocerebrosidase (GBA) gene are at high risk for cognitive impairment and approximately 10-17% of subjects undergoing DBS carry GBA mutations. There may be an interaction between STN-DBS, which also impairs cognitive function, and GBA, resulting in worsened cognitive function. This project will 1) determine the relationship between GBA mutation status and post-operative STN-DBS cognitive function, 2) broaden genotype-phenotype relationships of GBA mutation carriers and 3) provide scientific knowledge regarding the longitudinal cognitive effects of DBS in GBA mutation carriers through repeated neuropsychological testing.

DETAILED DESCRIPTION:
Parkinson disease (PD) is a neurodegenerative disease affecting at least 1 million people in the U.S. Each year, 9,000 PD patients undergo deep brain stimulator (DBS) placement into the subthalamic nucleus (STN-DBS), the most commonly used basal ganglia target. Despite motor improvement, up to 50% of patients have cognitive impairment after DBS. Cognitive impairment is associated with a 2-3 fold increase in mortality, progression to dementia, and nursing home placement. At present, subjects with cognitive impairment after DBS cannot be identified pre-operatively and the effects of DBS on cognitive function are not fully understood. A specific group of PD patients, carriers of mutations in the glucocerebrosidase (GBA) gene, are at particularly high risk for cognitive impairment. PD-GBA mutation carriers have dysfunction of the glucocerebrosidase (GCase) enzyme, resulting in more rapid accumulation and spread of Lewy bodies compared with non-mutation carriers. Clinically, PD-GBA mutation carriers have: (1) deficits in visual memory due to higher Lewy body burden in hippocampal and medial temporal regions, and (2) faster progression to dementia secondary to diffuse cortical Lewy body pathology. Approximately 10-17% of PD subjects with DBS carry GBA mutations, indicating that a substantial portion of the DBS population may be susceptible to cognitive problems. Importantly, STN-DBS itself can impair cognition through modulation of the striato-anterior cingulate cortex circuit, resulting in impulsivity and more errors when faced with tasks that rely on executive functions. Therefore, the central hypothesis is that PD-GBA mutation carriers have greater global cognitive decline after STN-DBS compared with PD-GBA mutation carriers without STN-DBS, and compared with non-mutation carriers with and without STN-DBS. This is a critical area of research because if an association between GBA and STN-DBS is detected, clinicians will be able to identify subjects at risk for worsened cognitive dysfunction through genetic testing and prevent harm by: (1) recommending that PD-GBA mutation carriers avoid STN-DBS, or (2) considering an alternative DBS target such as the globus pallidus interna (GPi) that may have less cognitive side effects. The following aims are proposed: Aim 1: Determine the longitudinal changes in global cognitive function in PD-GBA mutation carriers and non-mutation carriers with and without STN-DBS; Aim 2: Determine the specific pattern of cognitive dysfunction in PD-GBA mutation carriers and non-mutation carriers with and without STN-DBS; Aim 3: Determine the differential effects of DBS on cognitive function in the ON-stimulation state vs. OFF-stimulation state, comparing PD-GBA mutation and non-mutation carriers.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* onset of symptoms under age 60
* at least 5 years of disease
* with OR without deep brain stimulation

Exclusion Criteria:

* dementia

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease subjects with onset of symptoms under age 60 with moderate to advanced disease. Subjects can be with OR without deep brain stimulation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Mattis Dementia Rating Scale | 2 years
  scale to assess global cognition

SECONDARY OUTCOMES:
NIH toolbox cognition battery | 1 year
  iPAD based cognitive battery
Neuro-QoL | 2 years
  scale to assess quality of life
PROMIS | 2 years
  scale to assess quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Gian Pal, Principal Investigator — Rutgers University
Locations (1):
- Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pal GD, Hall D, Ouyang B, Phelps J, Alcalay R, Pauciulo MW, Nichols WC, Clark L, Mejia-Santana H, Blasucci L, Goetz CG, Comella C, Colcher A, Gan-Or Z, Rouleau GA, Marder K; Consortium on Risk for Early Onset Parkinson's Disease (CORE-PD) Investigators. Genetic and Clinical Predictors of Deep Brain Stimulation in Young-Onset Parkinson's Disease. Mov Disord Clin Pract. 2016 Sep-Oct;3(5):465-471. doi: 10.1002/mdc3.12309. Epub 2016 Jan 18. PMID 27709117